CLINICAL TRIAL: NCT00755846
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Comparison Study to Determine the Efficacy and Safety of SYR110322 in Patients With Type 2 Diabetes, Who Are Either Receiving No Current Treatment or Currently Treated With Diet and Exercise, Sulfonylurea, Metformin or a Combination of Sulfonylurea and Metformin
Brief Title: Safety and Efficacy Study of Alogliptin on Glycemic Control in Subjects With Type 2 Diabetes.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322-003; U1111-1113-8352 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Drug Therapy; Diabetes Mellitus, Type II; Type 2 Diabetes Mellitus; Hyperinsulinism; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Hyperinsulinism; Insulin Resistance | interventions — alogliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Alogliptin 6.25 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Alogliptin 12.5 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Alogliptin 25 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Alogliptin 50 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Alogliptin 100 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alogliptin — Alogliptin 6.25 mg, tablets, orally, once daily for up to 12 weeks
  Other Names: SYR-322; SYR110322
  Arms: Alogliptin 6.25 mg QD
Drug: Alogliptin — Alogliptin 12.5 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: SYR-322; SYR110322
  Arms: Alogliptin 12.5 mg QD
Drug: Alogliptin — Alogliptin 25 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: SYR-322; SYR110322
  Arms: Alogliptin 25 mg QD
Drug: Alogliptin — Alogliptin 50 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: SYR-322; SYR110322
  Arms: Alogliptin 50 mg QD
Drug: Alogliptin — Alogliptin 100 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: SYR-322; SYR110322
  Arms: Alogliptin 100 mg QD
Drug: Placebo — Alogliptin placebo-matching tablets, orally, once daily for up to 12 weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to determine the safety and efficacy of alogliptin, once daily (QD), compared to diet and exercise, sulfonylurea, metformin and a combination of sulfonylurea and metformin for treating subjects with type 2 diabetes.

DETAILED DESCRIPTION:
Of the approximately 19 million people in the United States who have been diagnosed with diabetes mellitus, 90% to 95% have type 2 diabetes mellitus. The prevalence of type 2 diabetes mellitus varies among racial and ethnic populations and has been shown to increase with age, obesity, family history, history of gestational diabetes, and physical inactivity. Over the next decade, a disproportionate increase in the elderly population will result in a marked increase in diabetic patients, placing an ever-increasing burden on families and the health care system.

In response to this problem, Takeda Global Research & Development Center, Inc. is developing SYR-322 (alogliptin), a selective, orally available inhibitor of the enzyme dipeptidyl peptidase IV. Dipeptidyl peptidase IV is thought to be primarily responsible for the in vivo degradation of 2 peptide hormones released in response to nutrient ingestion, namely glucagon-like peptide-1 and glucose-dependent insulinotropic peptide.

Individuals who want to participate in this study will be required to provide written informed consent. Study participation is anticipated to be about 14 Weeks. Multiple procedures will occur at each visit which may include blood collection, urine collection, vital signs including sitting and standing blood pressure and pulse, body height and weight, physical examinations and electrocardiograms.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes mellitus and were either receiving no current treatment or currently treated with a sulfonylurea, metformin, or a combination of a sulfonylurea and metformin but experiencing inadequate glycemic control. Subjects qualified as receiving no current treatment if 1 of the following conditions applied:

  * Subject was newly diagnosed (ie, had not received any treatment).
  * Subject was treated with diet and exercise alone for the 3 months prior to Screening
  * Subject had received <7 continuous days of any antidiabetic therapy within the 3 months prior to Screening.
  * Subject had a diagnosis of type 2 diabetes mellitus based on current American Diabetes Association criteria: fasting plasma glucose ≥126 mg/dL, oral glucose tolerance test at 2 hours after administration of the glucose load must have been ≥200 mg/dL, or symptoms of diabetes plus casual plasma glucose ≥200 mg/dL.
* Body mass index ≥23 kg/m2 and ≤40 kg/m2.
* Fasting C-peptide concentration ≥0.8 ng/mL.
* Glycosylated hemoglobin concentration between 6.8% and 11.0%.
* Fasting plasma glucose >126 mg/dL at Screening.
* No treatment within the 3 months prior to Screening with any other agents known to have effects on glucose (other than as described above, a sulfonylurea, metformin, or a combination of a sulfonylurea and metformin in subjects on antidiabetics), including but not limited to the following:

  * Other antidiabetic agents
  * Investigational antidiabetic agents
  * Niacin
  * Regular use of systemic glucocorticoids.
  * No treatment within the 3 months prior to Screening with weight-loss drugs
  * If taking other non-excluded medications, must have been on a stable dose of medication for at least 4 weeks.
* Diastolic blood pressure ≤110 mm Hg and a systolic pressure of ≤180 mm Hg.
* Female subjects could neither be pregnant (confirmed by laboratory testing) nor lactating, and if of childbearing potential must have been practicing adequate contraception.
* Able and willing to monitor their own blood glucose concentrations with a home glucose monitor.
* No major illness or debility that in the investigator's opinion prohibited the subject from completing the study.
* Hemoglobin ≥12 g/dL for males and ≥10 g/dL for females.
* Hepatic transaminase ≤2 x upper limit of normal.

Exclusion Criteria:

* History of cancer, other than squamous cell or basal cell carcinoma of the skin, that had not been in full remission for at least 1 year prior to Screening.
* History of proteinuria >1000 mg/day on a 12- or 24-hour urine collection OR a urine albumin/creatinine ratio >1000 μg/mg at Screening. If elevated, the subject was to be rescreened within 1 week.
* Serum creatinine ≥2.0 mg/dL.
* History of proliferative diabetic retinopathy OR any history of laser-treated retinopathy.
* History of treated peripheral or autonomic neuropathy.
* History of systolic dysfunction congestive heart failure.
* History of myocardial infarction within 1 year prior to Screening.
* History of ulcerative colitis or Crohn's disease.
* History of infection with hepatitis B, hepatitis C, or human immunodeficiency virus.
* History of a psychiatric disorder that would affect the subject's ability to participate in the study.
* History of anaphylactic reaction(s) to any drug.
* History of angioedema.
* History of alcohol or substance abuse within the last 2 years.
* History of any surgery that could potentially affect the absorption of the study drug.
* Receipt of any investigational drug within the preceding 30 days or a history of receipt of an investigational antidiabetic drug within the preceding 90 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2005-03; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda

REFERENCES:
- [Result] Pratley RE, McCall T, Fleck PR, Wilson CA, Mekki Q. Alogliptin use in elderly people: a pooled analysis from phase 2 and 3 studies. J Am Geriatr Soc. 2009 Nov;57(11):2011-9. doi: 10.1111/j.1532-5415.2009.02484.x. Epub 2009 Sep 30. PMID 19793357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 62 sites in Chile and the United States from 17 March 2005 to 10 June 2005.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus who were either receiving no current treatment or currently treated with diet and exercise, a sulfonylurea, metformin, or a combination of a sulfonylurea and metformin enrolled in once daily (QD) groups.
Groups:
- Placebo QD: Alogliptin placebo-matching tablets, orally, once daily for up to 12 weeks.
- Alogliptin 6.25 mg QD: Alogliptin 6.25 mg, tablets, orally, once daily for up to 12 weeks
- Alogliptin 12.5 mg QD: Alogliptin 12.5 mg, tablets, orally, once daily for up to 12 weeks.
- Alogliptin 25 mg QD: Alogliptin 25 mg, tablets, orally, once daily for up to 12 weeks.
- Alogliptin 50 mg QD: Alogliptin 50 mg, tablets, orally, once daily for up to 12 weeks.
- Alogliptin 100 mg QD: Alogliptin 100 mg, tablets, orally, once daily for up to 12 weeks.
Period: Overall Study
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Started | 43 | 44 | 44 | 45 | 44 | 45
Completed | 18 | 27 | 32 | 32 | 27 | 31
Not Completed | 25 | 17 | 12 | 13 | 17 | 14
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 3 | 2
Not completed — Protocol Violation | 1 | 1 | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0 | 4 | 2
Not completed — Withdrawal by Subject | 2 | 3 | 5 | 2 | 0 | 1
Not completed — Hyperglycemic Rescue | 21 | 7 | 5 | 8 | 8 | 7
Not completed — Physician Decision | 1 | 3 | 0 | 1 | 0 | 1
Not completed — Administrative Error | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Participant Non-compliance | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD | Total
Number analyzed (Participants) | 43 | 44 | 44 | 45 | 44 | 45 | 265
Age, Customized [Number; unit: participants]
  <65 years | 33 | 38 | 33 | 36 | 31 | 34 | 205
  ≥65 years | 10 | 6 | 11 | 9 | 13 | 11 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 22 | 17 | 26 | 25 | 139
  Male | 19 | 19 | 22 | 28 | 18 | 20 | 126

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Day 85.
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at day 85 or final visit and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Day 85.
Population: Randomized subjects who received at least 1 dose of study drug (Intent to Treat), and who had measurements at baseline and at Day 85. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Number analyzed (Participants) | 41 | 42 | 42 | 45 | 43 | 44
percentage of Glycosylated Hemoglobin | -0.01 (0.135) | -0.19 (0.121) | -0.54 (0.122) | -0.56 (0.117) | -0.44 (0.124) | -0.51 (0.119)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 6.25 mg QD vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD vs Alogliptin 50 mg QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in HbA1c. With at least 234 patients, a two-group t-test with a 0.05 two-sided significance has at least 98% power to detect a treatment difference (all active versus placebo) in HbA1c change from baseline as small as 0.55%, assuming a common standard deviation of 0.7%; Test type: Superiority or Other; p = 0.001, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and body mass index (BMI), diabetes duration and baseline HbA1c as covariates; Mean Difference (Final Values) = -0.43, Standard Error of Mean 0.135 — Negative mean treatment difference indicates larger decrease from baseline (more negative change from baseline) in the alogliptin arm compared to the placebo arm
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in HbA1c. With at least 234 patients, a two-group t-test with a 0.05 two-sided significance level has 90% power to detect a treatment difference (each active dose versus placebo) in HbA1c change from baseline as small as 0.55%, assuming a common standard deviation of 0.7%; Test type: Superiority or Other; p = 0.004, ANCOVA — A step-down sequential approach was used to test the hypothesis that the treatment coefficient in the model is 0 for each of the five individual active treatment groups vs. placebo; Treatment and prior antidiabetic treatment as class effects and BMI, diabetes duration, and baseline HbA1c as covariates; Mean Difference (Final Values) = -0.50, Standard Error of Mean 0.171 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo QD vs Alogliptin 50 mg QD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.017, ANCOVA — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 2]; Mean Difference (Net) = -0.42, Standard Error of Mean 0.176 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo QD vs Alogliptin 25 mg QD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.55, Standard Error of Mean 0.170 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.52, Standard Error of Mean 0.174 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo QD vs Alogliptin 6.25 mg QD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.307, ANCOVA — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.18, Standard Error of Mean 0.173 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin at Day 43.
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at day 43 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Day 43.
Population: Randomized subjects who received at least 1 dose of study drug (Intent to treat), and who had measurements at baseline and at Day 43. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Number analyzed (Participants) | 41 | 42 | 42 | 44 | 43 | 44
percentage of Glycosylated Hemoglobin | 0.02 (0.097) | -0.12 (0.095) | -0.35 (0.096) | -0.36 (0.093) | -0.32 (0.097) | -0.31 (0.094)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 6.25 mg QD vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD vs Alogliptin 50 mg QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in HbA1c. With at least 234 patients, a two-group t-test with a 0.05 two-sided significance level has at least 98% power to detect a treatment difference (all active versus placebo) in HbA1c change from baseline as small as 0.55%, assuming a common standard deviation of 0.7%; Test type: Superiority or Other; p = 0.004, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.31, Standard Error of Mean 0.106 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 100 mg QD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.017, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.32, Standard Error of Mean 0.134 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo QD vs Alogliptin 50 mg QD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.016, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.34, Standard Error of Mean 0.138 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo QD vs Alogliptin 25 mg QD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.005, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.38, Standard Error of Mean 0.134 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.008, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.37, Standard Error of Mean 0.137 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo QD vs Alogliptin 6.25 mg QD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.321, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.14, Standard Error of Mean 0.136 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Day 43).
Description: The change between the value of fasting plasma glucose collected at day 43 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Day 43
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Number analyzed (Participants) | 41 | 42 | 42 | 45 | 43 | 44
mg/dL | 4.9 (6.09) | -7.3 (6.00) | -11.5 (6.02) | -24.5 (5.80) | -17.9 (6.10) | -25.6 (5.88)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 6.25 mg QD vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD vs Alogliptin 50 mg QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in fasting plasma glucose (FPG). The treatment effect was evaluated as a contrast of all doses of alogliptin versus placebo and was evaluated inferentially with a 2-sided t-test at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and body mass index (BMI), diabetes duration, and baseline FPG as covariates; Mean Difference (Final Values) = -22.2, Standard Error of Mean 6.65 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in FPG. The treatment effect was evaluated as a contrast of each dose of alogliptin versus placebo and was evaluated inferentially with a 2-sided t-test at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and BMI, diabetes duration, and baseline FPG as covariates; Mean Difference (Final Values) = -30.5, Standard Error of Mean 8.40 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo QD vs Alogliptin 50 mg QD; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.009, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and BMI, diabetes duration, and baseline FPG as covariates; Mean Difference (Final Values) = -22.8, Standard Error of Mean 8.68 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo QD vs Alogliptin 25 mg QD; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and BMI, diabetes duration, and baseline FPG as covariates; Mean Difference (Final Values) = -29.4, Standard Error of Mean 8.38 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.057, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and BMI, diabetes duration, and baseline FPG as covariates; Mean Difference (Final Values) = -16.4, Standard Error of Mean 8.57 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo QD vs Alogliptin 6.25 mg QD; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.156, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and BMI, diabetes duration, and baseline FPG as covariates; Mean Difference (Final Values) = -12.2, Standard Error of Mean 8.56 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Day 85).
Description: The change between the value of fasting plasma glucose collected at day 85 or final visit and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Day 85.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Number analyzed (Participants) | 41 | 42 | 42 | 45 | 43 | 44
mg/dL | 8.5 (6.45) | -7.8 (6.36) | -5.1 (6.39) | -27.0 (6.14) | -16.1 (6.47) | -20.9 (6.23)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 6.25 mg QD vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD vs Alogliptin 50 mg QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between all doses of alogliptin and placebo arms in change from baseline in FPG. The treatment effect was evaluated as a contrast of all doses of alogliptin versus placebo and was evaluated inferentially with a 2-sided t-test at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and BMI, diabetes duration, and baseline FPG as covariates; Mean Difference (Final Values) = -23.9, Standard Error of Mean 7.05 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 100 mg QD; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.001, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and BMI, diabetes duration, and baseline FPG as covariates; Mean Difference (Final Values) = -29.4, Standard Error of Mean 8.91 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo QD vs Alogliptin 50 mg QD; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.008, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and BMI, diabetes duration, and baseline FPG as covariates; Mean Difference (Final Values) = -24.6, Standard Error of Mean 9.20 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo QD vs Alogliptin 25 mg QD; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and body mass index, diabetes duration, and baseline HbA1c as covariates; Mean Difference (Final Values) = -35.5, Standard Error of Mean 8.88 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.136, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -13.6, Standard Error of Mean 9.09 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo QD vs Alogliptin 6.25 mg QD; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.073, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -16.3, Standard Error of Mean 9.07 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline in Fasting Fructosamine (Day 43).
Description: The change between the value of fasting fructosamine collected at day 43 and fasting fructosamine collected at baseline.
Time Frame: Baseline and Day 43.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Number analyzed (Participants) | 39 | 41 | 42 | 43 | 39 | 43
mg/dL | 7.6 (5.35) | -4.2 (5.16) | -13.1 (5.12) | -14.5 (5.05) | -16.3 (5.47) | -11.7 (5.09)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 6.25 mg QD vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD vs Alogliptin 50 mg QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in fasting fructosamine. The treatment effect will be evaluated as a contrast of all doses of alogliptin versus placebo and was evaluated inferentially with a 2-sided t-test at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and BMI, diabetes duration, and baseline fasting fructosamine as covariates; Mean Difference (Final Values) = -19.5, Standard Error of Mean 5.85 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in fasting fructosamine. The treatment effect was evaluated as a contrast of each dose of alogliptin versus placebo and was evaluated inferentially with a 2-sided t-test at the 0.05 significance level; Test type: Superiority or Other; p = 0.010, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -19.2, Standard Error of Mean 7.37 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo QD vs Alogliptin 50 mg QD; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.002, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -23.8, Standard Error of Mean 7.71 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo QD vs Alogliptin 25 mg QD; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.003, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -22.1, Standard Error of Mean 7.33 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.006, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -20.7, Standard Error of Mean 7.44 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo QD vs Alogliptin 6.25 mg QD; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.117, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -11.7, Standard Error of Mean 7.45 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline in Fasting Fructosamine (Day 85).
Description: The change between the value of fasting fructosamine collected at day 85 or final visit and fasting fructosamine collected at baseline.
Time Frame: Baseline and Day 85.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Number analyzed (Participants) | 41 | 42 | 42 | 45 | 40 | 44
mg/dL | 7.7 (6.03) | 0.2 (5.91) | -9.8 (5.93) | -16.4 (5.71) | -12.4 (6.25) | -4.8 (5.82)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 6.25 mg QD vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD vs Alogliptin 50 mg QD vs Alogliptin 100 mg QD; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.014, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -16.3, Standard Error of Mean 6.60 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 100 mg QD; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.136, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -12.5, Standard Error of Mean 8.35 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo QD vs Alogliptin 50 mg QD; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.022, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -20.1, Standard Error of Mean 8.73 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo QD vs Alogliptin 25 mg QD; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.004, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -24.1, Standard Error of Mean 8.26 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Alogliptin 12.5 mg QD; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.040, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -17.5, Standard Error of Mean 8.48 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo QD vs Alogliptin 6.25 mg QD; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.378, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -7.5, Standard Error of Mean 8.47 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in Total Cholesterol (Day 43).
Description: The change between the value of cholesterol collected at day 43 and cholesterol collected at baseline.
Time Frame: Baseline and Day 43
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Number analyzed (Participants) | 40 | 41 | 42 | 43 | 39 | 42
mg/dL | -11.1 (4.91) | -9.7 (4.85) | -9.6 (4.77) | -9.8 (4.71) | -12.0 (5.11) | -4.7 (4.80)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 6.25 mg QD vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD vs Alogliptin 50 mg QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in total cholesterol. The treatment effect will be evaluated as a contrast of all doses of alogliptin versus placebo and was evaluated inferentially with a 2-sided t-test at the 0.05 significance level; Test type: Superiority or Other; p = 0.718, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and BMI, diabetes duration, and baseline total cholesterol as covariates; Mean Difference (Final Values) = 1.9, Standard Error of Mean 5.37 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in total cholesterol. The treatment effect was evaluated as a contrast of each dose of alogliptin versus placebo and was evaluated inferentially with a 2-sided t-test at the 0.05 significance level; Test type: Superiority or Other; p = 0.346, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 6.4, Standard Error of Mean 6.80 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo QD vs Alogliptin 50 mg QD; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.901, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.9, Standard Error of Mean 7.13 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo QD vs Alogliptin 25 mg QD; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.851, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 1.3, Standard Error of Mean 6.79 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.825, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 1.5, Standard Error of Mean 6.86 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo QD vs Alogliptin 6.25 mg QD; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.843, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 1.4, Standard Error of Mean 6.94 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline in Total Cholesterol (Day 85).
Description: The change between the value of cholesterol collected at day 85 or final visit and cholesterol collected at baseline.
Time Frame: Baseline and Day 85.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Number analyzed (Participants) | 41 | 42 | 42 | 45 | 40 | 44
mg/dL | -15.1 (4.46) | -9.0 (4.41) | -4.8 (4.39) | -8.7 (4.24) | -7.7 (4.64) | -0.4 (4.31)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 6.25 mg QD vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD vs Alogliptin 50 mg QD vs Alogliptin 100 mg QD; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.069, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 8.9, Standard Error of Mean 4.88 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 100 mg QD; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.018, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 14.6, Standard Error of Mean 6.14 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo QD vs Alogliptin 50 mg QD; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.258, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 7.3, Standard Error of Mean 6.47 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo QD vs Alogliptin 25 mg QD; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.299, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 6.4, Standard Error of Mean 6.13 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.103, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 10.3, Standard Error of Mean 6.27 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo QD vs Alogliptin 6.25 mg QD; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.340, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 6.0, Standard Error of Mean 6.32 — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change From Baseline in High-Density Lipoprotein Cholesterol (Day 43).
Description: The change between high-density lipoprotein cholesterol collected at day 43 and high-density lipoprotein cholesterol collected at baseline.
Time Frame: Baseline and Day 43.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Number analyzed (Participants) | 40 | 41 | 42 | 43 | 39 | 42
mg/dL | -1.4 (0.76) | -0.6 (0.75) | -2.0 (0.74) | -2.4 (0.73) | -2.8 (0.80) | -1.1 (0.74)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 6.25 mg QD vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD vs Alogliptin 50 mg QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in HDL cholesterol. The treatment effect will be evaluated as a contrast of all doses of alogliptin versus placebo and was evaluated inferentially with a 2-sided t-test at the 0.05 significance level; Test type: Superiority or Other; p = 0.689, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and BMI, diabetes duration, and baseline HDL cholesterol as covariates; Mean Difference (Final Values) = -0.3, Standard Error of Mean 0.83 — Positive mean treatment difference indicates larger increase from baseline (more positive change from baseline) in the alogliptin arm compared to the placebo arm
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in HDL cholesterol. The treatment effect was evaluated as a contrast of each dose of alogliptin versus placebo and was evaluated inferentially with a 2-sided t-test at the 0.05 significance level; Test type: Superiority or Other; p = 0.742, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.3, Standard Error of Mean 1.05 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Placebo QD vs Alogliptin 50 mg QD; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.220, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -1.4, Standard Error of Mean 1.11 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Placebo QD vs Alogliptin 25 mg QD; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.348, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -1.0, Standard Error of Mean 1.05 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.627, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.5, Standard Error of Mean 1.06 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Placebo QD vs Alogliptin 6.25 mg QD; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.418, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.9, Standard Error of Mean 1.06 — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Change From Baseline in High-Density Lipoprotein Cholesterol (Day 85).
Description: The change between high-density lipoprotein cholesterol collected at day 85 or final visit and high-density lipoprotein cholesterol collected at baseline.
Time Frame: Baseline and Day 85.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Number analyzed (Participants) | 41 | 42 | 42 | 45 | 40 | 44
mg/dL | -1.9 (0.87) | -0.7 (0.86) | -2.3 (0.85) | -2.5 (0.83) | -2.0 (0.92) | 0.4 (0.84)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 6.25 mg QD vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD vs Alogliptin 50 mg QD vs Alogliptin 100 mg QD; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.617, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.5, Standard Error of Mean 0.95 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 100 mg QD; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.052, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 2.3, Standard Error of Mean 1.20 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Placebo QD vs Alogliptin 50 mg QD; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.906, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.2, Standard Error of Mean 1.28 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Placebo QD vs Alogliptin 25 mg QD; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.628, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.6, Standard Error of Mean 1.19 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.749, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.4, Standard Error of Mean 1.22 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Placebo QD vs Alogliptin 6.25 mg QD; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.340, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.2, Standard Error of Mean 1.22 — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Change From Baseline in Low-Density Lipoprotein Cholesterol (Day 43).
Description: The change between low-density lipoprotein cholesterol collected at day 43 and low-density lipoprotein cholesterol collected at baseline.
Time Frame: Baseline and Day 43.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Number analyzed (Participants) | 35 | 38 | 39 | 40 | 36 | 37
mg/dL | -8.9 (3.97) | -3.8 (3.79) | -6.4 (3.72) | -1.5 (3.69) | -9.9 (4.01) | 0.8 (3.84)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 6.25 mg QD vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD vs Alogliptin 50 mg QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in LDL cholesterol. The treatment effect will be evaluated as a contrast of all doses of alogliptin versus placebo and was evaluated inferentially with a 2-sided t-test at the 0.05 significance level; Test type: Superiority or Other; p = 0.269, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and BMI, diabetes duration, and baseline LDL cholesterol as covariates; Mean Difference (Final Values) = 4.8, Standard Error of Mean 4.31 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in LDL cholesterol. The treatment effect was evaluated as a contrast of each dose of alogliptin versus placebo and was evaluated inferentially with a 2-sided t-test at the 0.05 significance level; Test type: Superiority or Other; p = 0.076, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 9.7, Standard Error of Mean 5.46 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo QD vs Alogliptin 50 mg QD; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.867, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.9, Standard Error of Mean 5.66 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo QD vs Alogliptin 25 mg QD; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.169, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 7.4, Standard Error of Mean 5.40 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.645, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 2.5, Standard Error of Mean 5.45 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo QD vs Alogliptin 6.25 mg QD; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.351, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 5.2, Standard Error of Mean 5.51 — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Change From Baseline in Low-Density Lipoprotein Cholesterol (Day 85).
Description: The change between low-density lipoprotein cholesterol collected at day 85 or final visit and low-density lipoprotein cholesterol collected at baseline.
Time Frame: Baseline and Day 85.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Number analyzed (Participants) | 36 | 39 | 39 | 43 | 38 | 40
mg/dL | -13.6 (3.72) | -2.6 (3.55) | -2.7 (3.54) | -0.6 (3.38) | -5.0 (3.70) | 4.0 (3.50)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 6.25 mg QD vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD vs Alogliptin 50 mg QD vs Alogliptin 100 mg QD; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.003, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 12.3, Standard Error of Mean 4.03 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 100 mg QD; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 17.6, Standard Error of Mean 5.06 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo QD vs Alogliptin 50 mg QD; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.103, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 8.6, Standard Error of Mean 5.26 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo QD vs Alogliptin 25 mg QD; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.009, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 13.0, Standard Error of Mean 4.98 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.034, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 11.0, Standard Error of Mean 5.14 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo QD vs Alogliptin 6.25 mg QD; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.033, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 11.1, Standard Error of Mean 5.16 — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Change From Baseline in Triglycerides (Day 43).
Description: The change between triglycerides collected at day 43 and triglycerides collected at baseline.
Time Frame: Baseline and Day 43.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Number analyzed (Participants) | 40 | 41 | 42 | 43 | 39 | 42
mg/dL | -18.7 (15.69) | -28.0 (15.43) | -10.1 (15.28) | -27.7 (15.10) | -7.2 (16.33) | -31.5 (15.48)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 6.25 mg QD vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD vs Alogliptin 50 mg QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in triglycerides. The treatment effect will be evaluated as a contrast of all doses of alogliptin versus placebo and was evaluated inferentially with a 2-sided t-test at the 0.05 significance level; Test type: Superiority or Other; p = 0.897, ANCOVA — No multiplicity adjustments; Treatment and prior antidiabetic treatment as class effects and BMI, diabetes duration, and baseline triglycerides as covariates; Mean Difference (Final Values) = -2.2, Standard Error of Mean 17.17 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 100 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in triglycerides. The treatment effect was evaluated as a contrast of each dose of alogliptin versus placebo and was evaluated inferentially with a 2-sided t-test at the 0.05 significance level; Test type: Superiority or Other; p = 0.557, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 13, analysis 1]; Mean Difference (Final Values) = -12.8, Standard Error of Mean 21.85 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo QD vs Alogliptin 50 mg QD; [analysis description as in outcome 13, analysis 2]; Test type: Superiority or Other; p = 0.616, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 13, analysis 1]; Mean Difference (Final Values) = 11.5, Standard Error of Mean 22.85 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo QD vs Alogliptin 25 mg QD; [analysis description as in outcome 13, analysis 2]; Test type: Superiority or Other; p = 0.679, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 13, analysis 1]; Mean Difference (Final Values) = -9.0, Standard Error of Mean 21.73 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; [analysis description as in outcome 13, analysis 2]; Test type: Superiority or Other; p = 0.697, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 13, analysis 1]; Mean Difference (Final Values) = 8.5, Standard Error of Mean 21.94 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo QD vs Alogliptin 6.25 mg QD; [analysis description as in outcome 13, analysis 2]; Test type: Superiority or Other; p = 0.672, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 13, analysis 1]; Mean Difference (Final Values) = -9.4, Standard Error of Mean 22.03 — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Change From Baseline in Triglycerides (Day 85).
Description: The change between triglycerides collected at day 85 or final visit and triglycerides collected at baseline.
Time Frame: Baseline and Day 85.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Number analyzed (Participants) | 41 | 42 | 42 | 45 | 40 | 44
mg/dL | -13.9 (14.98) | -26.4 (14.75) | 9.2 (14.77) | -32.9 (14.27) | -14.4 (15.58) | -24.9 (14.59)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 6.25 mg QD vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD vs Alogliptin 50 mg QD vs Alogliptin 100 mg QD; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.809, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 13, analysis 1]; Mean Difference (Final Values) = -4.0, Standard Error of Mean 16.37 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 100 mg QD; [analysis description as in outcome 13, analysis 2]; Test type: Superiority or Other; p = 0.597, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 13, analysis 1]; Mean Difference (Final Values) = -11.0, Standard Error of Mean 20.74 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo QD vs Alogliptin 50 mg QD; [analysis description as in outcome 13, analysis 2]; Test type: Superiority or Other; p = 0.982, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 13, analysis 1]; Mean Difference (Final Values) = -0.5, Standard Error of Mean 21.77 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo QD vs Alogliptin 25 mg QD; [analysis description as in outcome 13, analysis 2]; Test type: Superiority or Other; p = 0.358, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 13, analysis 1]; Mean Difference (Final Values) = -19.0, Standard Error of Mean 20.62 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; [analysis description as in outcome 13, analysis 2]; Test type: Superiority or Other; p = 0.274, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 13, analysis 1]; Mean Difference (Final Values) = 23.1, Standard Error of Mean 21.06 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo QD vs Alogliptin 6.25 mg QD; [analysis description as in outcome 13, analysis 2]; Test type: Superiority or Other; p = 0.554, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 13, analysis 1]; Mean Difference (Final Values) = -12.5, Standard Error of Mean 21.06 — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Mean Percent Incidence of Marked Hyperglycemia (Fasting Plasma Glucose ≥ 200 mg/dL).
Description: The incidence of marked hyperglycemia occurring in participants with a fasting plasma glucose value greater than or equal to 200 mg per dL during study. Overall mean obtained by weighting the hyperglycemia percent incidence values at each time point by number of days in between visits. Mean percent incidence of marked hyperglycemia at each time point is the percent of self-monitored blood glucose measurements greater than or equal to 200 mg per dL, calculated per participant and then averaged across population.
Time Frame: 85 Days.
Population: Randomized participants who received at least 1 dose of study drug (Intent to Treat), and who had at least 1 fasting plasma glucose measurement after baseline.
  Note: Mean percent incidence of marked hyperglycemia was only summarized by treatment group using descriptive statistics.
Measure: Mean (Standard Deviation); unit: percent incidence
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Number analyzed (Participants) | 41 | 42 | 42 | 45 | 43 | 44
percent incidence | 54.0 (34.95) | 34.7 (33.43) | 25.8 (26.92) | 28.1 (25.94) | 30.4 (30.32) | 30.6 (29.92)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days after the last dose of double-blind drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo QD | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Alogliptin 100 mg QD
Serious Adverse Events (participants affected / at risk) | 2/41 | 1/42 | 0/44 | 1/45 | 0/43 | 0/44
Other Adverse Events (participants affected / at risk) | 14/41 | 12/42 | 18/44 | 19/45 | 15/43 | 22/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD (N=41) | Alogliptin 6.25 mg QD (N=42) | Alogliptin 12.5 mg QD (N=44) | Alogliptin 25 mg QD (N=45) | Alogliptin 50 mg QD (N=43) | Alogliptin 100 mg QD (N=44)
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Noncardiac chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD (N=41) | Alogliptin 6.25 mg QD (N=42) | Alogliptin 12.5 mg QD (N=44) | Alogliptin 25 mg QD (N=45) | Alogliptin 50 mg QD (N=43) | Alogliptin 100 mg QD (N=44)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 3 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 3 | 1 | 1
Fatigue (General disorders) | 2 | 0 | 1 | 0 | 2 | 3
Fungal infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 0 | 4 | 3 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 2 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 1 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 4 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 1
Urinary tract infection (Infections and infestations) | 4 | 3 | 1 | 3 | 3 | 4
Vision blurred (Eye disorders) | 0 | 1 | 1 | 2 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.